CLINICAL TRIAL: NCT05788185
Title: Phase 1b, Randomized, Open-label Study to Evaluate the Safety, Tolerability, and Immunogenicity of RVM-V001 Only, RVM-V002 Only, or RVM V001 + RVM V002 (Co Administered as Separate Injections) in Healthy Adults Previously Vaccinated With an Inactivated Virus or mRNA-based COVID-19 Vaccine in Singapore
Brief Title: Safety & Immunogenicity of RVM-V001/RVM-V002 or RVMV001+RVMV002 (Co Administered as Separate Injections) in Healthy Individuals
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Changes in COVID-19 pandemic landscape
Sponsor: RVAC Medicines (US), Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RV003
Record Dates: First submitted 2023-02-21; First posted 2023-03-28 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Infectious Disease; COVID-19
MeSH Terms: conditions — Communicable Diseases; COVID-19 | interventions — RVM-V001 COVID-19 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- RVM-V001 30 µg -BNT162b2 subjects (Experimental): RVM-V001-30 µg administered as a single dose of by intramuscular injection on Day 1 on BNT162b2 subjects
  Interventions: Biological: RVM-V001 30 µg
- RVM-V002 30 µg -BNT162b2 subjects (Experimental): RVM-V001-30 µg administered as a single dose of by intramuscular injection on Day 1 on BNT162b2 subjects
  Interventions: Biological: RVM-V002 30 µg
- RVM-V001 (15 µg) + RVM-V002 (15 µg) co-administration -BNT162b2 subjects (Experimental): RVM-V001 (15 µg) + RVM-V002 (15 µg) co-administration; a single dose of RVM-V001 in the left arm deltoid muscle and then followed immediately with a single dose of RVM-V002 in the right arm deltoid muscle on Day 1 on BNT162b2 subjects
  Interventions: Biological: RVM-V001 (15 µg) + RVM-V002 (15 µg) co-administration
- RVM-V001 30 µg (Experimental): RVM-V001-30 µg administered as a single dose of by intramuscular injection on Day 1 on BBIBP-CorV or CoronaVac subjects
  Interventions: Biological: RVM-V001 30 µg
- RVM-V002-30 µg (Experimental): RVM-V002-30 µg administered as a single dose of by intramuscular injection on Day 1 on BBIBP-CorV or CoronaVac subjects
  Interventions: Biological: RVM-V002 30 µg
- RVM-V001 (15 µg) + RVM-V002 (15 µg) co-administration (Experimental): RVM-V001 (15 µg) + RVM-V002 (15 µg) co-administration; a single dose of RVM-V001 in the left arm deltoid muscle and then followed immediately with a single dose of RVM-V002 in the right arm deltoid muscle on Day 1 on BBIBP-CorV or CoronaVac subjects
  Interventions: Biological: RVM-V001 (15 µg) + RVM-V002 (15 µg) co-administration

INTERVENTIONS:
Biological: RVM-V001 30 µg — For BNT162b2 subjects
  Arms: RVM-V001 30 µg -BNT162b2 subjects
Biological: RVM-V002 30 µg — For BNT162b2 subjects
  Arms: RVM-V002 30 µg -BNT162b2 subjects
Biological: RVM-V001 (15 µg) + RVM-V002 (15 µg) co-administration — For BNT162b2 subjects
  Arms: RVM-V001 (15 µg) + RVM-V002 (15 µg) co-administration -BNT162b2 subjects
Biological: RVM-V001 30 µg — For BBIBP-CorV or CoronaVac subjects
  Arms: RVM-V001 30 µg
Biological: RVM-V002 30 µg — For BBIBP-CorV or CoronaVac subjects
  Arms: RVM-V002-30 µg
Biological: RVM-V001 (15 µg) + RVM-V002 (15 µg) co-administration — For BBIBP-CorV or CoronaVac subjects
  Arms: RVM-V001 (15 µg) + RVM-V002 (15 µg) co-administration

SUMMARY:
Phase 1b, randomized, open-label, study to evaluate the safety, tolerability, and immunogenicity of RVM-V001 only, RVM-V002 only, or RVM V001 + RVM V002 (Co administered as Separate Injections) in healthy adults. The study will be conducted at one site in Singapore.

DETAILED DESCRIPTION:
A total of 48 healthy men and non-pregnant women aged 21 years and older will be stratified by prior vaccination. Twenty-four subjects who have received a 3 dose primary vaccination series, with or without 1 booster dose, of an approved inactivated virus vaccine (BBIBP-CorV or CoronaVac) will be randomized at a 1:1:1 ratio to receive RVM V001 (30 µg) only, RVM V002 (30 µg) only, or RVM-V001 (15 µg) + RVM V002 (15ug).

An additional 24 subjects who have received 3 doses (primary vaccination series and 1 booster dose) of an mRNA vaccine (BNT162b2) will be randomized at 1:1:1 ratio to receive RVM-V001 (30 µg) only, RVM V002 (30 µg) only, or RVM-V001 (15 µg ) + RVM V002 (15 µg ). The last dose of the prior vaccination should have been administered at least 6 months prior to enrolment in this study. For administration of RVM V001 only or RVM V002 only, subjects will receive a single dose of RVM-V001 or RMV-V002 vaccine on Day 1 via intramuscular (IM) injection into deltoid muscle, preferably of the non-dominant arm.

For the RVM V001 + RVM V002 administration, subjects will receive a single dose of RVM-V001 in the left arm deltoid muscle and then followed immediately with a single dose of RVM-V002 in the right arm deltoid muscle.

ELIGIBILITY:
Inclusion Criteria:

* Male and female healthy volunteers.
* Aged 21 years and older on Day 1
* Judged by the investigator to be healthy based on medical history, physical examination, and vital signs evaluation at Screening visit.
* Able to provide informed consent form.
* Able and willing to comply with all study procedures over follow-up period of approximately 6 months.
* Have documented completion of a 2-dose primary vaccination series and 1 booster vaccination with BNT162b2 OR a 3-dose primary vaccination series, with or without 1 booster dose, with an approved inactivated virus vaccine (BBIBP-CorV or CoronaVac). The last dose in all cases should have been administered at least 6 months prior to enrolment in this study.
* For female subjects with childbearing potential: must agree to avoid pregnancy from 21 days prior to Day 1 until at least 90 days after the last study vaccination. Women physically capable of pregnancy (not sterilized and still menstruating or within 1 year of the last menses if menopausal) in sexual relationships with men must use an acceptable method of avoiding pregnancy during this period.

Exclusion Criteria:

* Received any COVID-19 vaccine other than BNT162b2, BBIBP-CorV, or CoronaVac.
* Received more than 3 doses of BNT162b2 or more than 4 doses of BBIBP-CorV or CoronaVac.
* Women who are pregnant or breastfeeding or intending to become pregnant; mend who will father children within the projected duration of the trial.
* Positive serology test results for hepatitis C virus antibody, human immunodeficiency virus antibody, or hepatitis B viral surface antigen at Screening.
* Is currently participating in or has participated in a study with an investigational product within 30 days preceding Day 1.
* History of severe allergic reactions (eg, acute anaphylaxis, urticaria, skin eczema, dyspnoea, angioneurotic oedema) or other significant adverse reactions to COVID19 vaccines; allergy to known composition of RVM-001 and RVM-002.
* History of coagulation dysfunction (eg, coagulation factor deficiency, coagulation disease).
* Vaccinated with live attenuated vaccine within 1 month, or any other vaccine within 14 days, of Day 1 vaccination.
* Received systemic immunosuppressants within 4 months prior to vaccination or an anticipated need for immunosuppressants at any time during the study. Topical or inhaled treatment is allowed if not used within 14 days prior to Day 1 vaccination.
* Received blood products within 3 months prior to Day 1 vaccination.
* History of alcohol or drug abuse within 3 years prior to Day 1 vaccination.
* Fever (temperature > 37.5°C), dry cough, fatigue, nasal obstruction, runny nose, sore throat, myalgia, diarrhoea, shortness of breath, or dyspnoea on the day of vaccination.
* Any condition that, in the opinion of the investigator, would pose a health risk to the subject if enrolled, could interfere with the evaluation of the study vaccine, or interfere with interpretation of the study results (including neurologic or psychiatric conditions deemed likely to impair the quality of safety reporting).

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
Safety in terms of solicited adverse events | Day 1 to Day 7 inclusive
  Number of subjects with solicited adverse events
Safety in terms of solicited systemic adverse events | Day 1 to Day 7 inclusive
  Number of subjects with solicited systemic adverse events
Safety in terms of unsolicited adverse events | Day 1 to Day 28 inclusive
  Number of subjects with unsolicited adverse events
Safety in terms of SAEs, SUSARs, MAAEs and AESIs | Day 1 to Day 180 post dose
  Number of subjects with SAEs, SUSARs, MAAEs and AESIs
Safety in terms of laboratory-based AEs | Day 1 to Day 180 post dose
  Changes in safety laboratory parameters from baseline by the Food and Drug Administration (FDA) toxicity grading scale.

SECONDARY OUTCOMES:
Immunogenicity in terms of Nab | Days 1,8,15,29 and 180
  GMT of neutralizing antibody (pseudoviral neutralization assay) against Wuhan strain and BA.1 subvariant
GMT of neutralizing antibody (pseudoviral neutralization assay) against Variants of Immunogenicity in terms of Nab | Days 1,8,15,29 and 180
  GMT of neutralizing antibody (pseudoviral neutralization assay) against Variants of concerns of SARS-CoV-2
Immunogenicity in terms of Humoral immune response by ELISA | Days 1,8,15,29 and 180
  GMT of serum binding antibodies (IgG) by ELISA
Seroresponse rate for neutralizing antibody | Days 8,15,29 and 180
  SRR percentage of subjects with ≥4-fold increase of antibody titer over baseline
Seroresponse rate for binding antibodies (IgG) by ELISA | Days 8,15,29 and 180
  SRR percentage of subjects with ≥4-fold increase of antibody titer over baseline
Geometric Mean Fold Rise (GMFR) of SARS-CoV-2 Neutralizing Antibody | Days 8,15,29 and 180
Geometric Mean Fold Rise (GMFR) of binding antibodies (IgG) by ELISA | Days 8,15,29 and 180

CONTACTS AND LOCATIONS:
Locations (1):
- P.H. Feng Research Centre, NCID,TTSH, Singapore, Singapore